CLINICAL TRIAL: NCT06875219
Title: An Observational Study to Evaluate Long- Term Safety and Efficacy of Luspatercept in Subjects with Transfusion Dependent Who Received the First Dose of Luspatercept After Its Introduction in the Clinical Practice
Brief Title: To Evaluate Long- Term Safety and Efficacy of Luspatercept
Acronym: LUSPAREAL001
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione per la Ricerca sulle Anemie ed Emoglobinopatie in Italia (Other)
Responsible Party: Sponsor
Other Study IDs: LUSPAREAL001
Record Dates: First submitted 2025-02-25; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia | interventions — luspatercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Luspatercept (ACE-536) — Luspatercept (ACE-536)

SUMMARY:
An observational study to evaluate long-term safety and efficacy of luspatercept in subjects with transfusion dependent who received the first dose of luspatercept after its introduction in the clinical practice

DETAILED DESCRIPTION:
Luspatercept represents the first and only erythroid maturation agent (EMA) approved by the European Commission (EC) and the Food and Drug Administration (FDA) capable of enhancing advanced erythrocyte maturation. The efficacy of luspatercept was demonstrated in the phase III clinical trial called "BELIEVE." With market authorization, the drug is used in less selected patients with potentially more complex medical histories than those enrolled in the registration study. In addition, it is now also possible to prescribe the drug in patients with blood consumption at baseline between 20 and 24 blood units in the 24 weeks before the drug was prescribed, who could not be included in the "BELIEVE" study. Gathering data on the clinical characteristics of patients who are prescribed luspatercept in normal clinical practice, and of safety and efficacy in this setting, is essential to enrich the available information on this new therapy.

ELIGIBILITY:
Inclusion criteria:

Subjects who received at least one dose of luspatercept after its introduction in the clinical practice

Exclusion Criteria:

* Subjects who received luspatercept after participating in the "compassionate" use program
* Subjects unwilling to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (male and female), living or deceased patients with transfusion-dependent beta thalassemia who received the first dose of luspatercept after its introduction in the clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2026-02-24 (Estimated)

PRIMARY OUTCOMES:
Safety of luspatercept - Number of participants with treatment-related adverse events as assessed by CTCAE v4.0" | 52 WEEK
  - To evaluate safety of luspatercept in subjects with transfusion-dependent beta thalassemia who received the first dose of luspatercept after its introduction in the clinical practice
Tolerability of luspatercept - Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 52 WEEK
  - To evaluate tolerability of luspatercept in subjects with transfusion-dependent beta thalassemia who received the first dose of luspatercept after its introduction in the clinical practice
Efficacy of luspatercept - Number of subjects who showed a ≥ 33% reduction from baseline in the number of transfused blood units during any 12-week interval period of luspatercept treatment | 12 weeks
  - To evaluate efficacy of luspatercept in subjects with transfusion-dependent beta thalassemia who received the first dose of luspatercept after its introduction in the clinical practice

SECONDARY OUTCOMES:
safety of luspatercept - Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 52 weeks
  - To evaluate safety of luspatercept in subjects with transfusion-dependent beta thalassemia with baseline transfusion needs and comorbidities that were exclusion criteria in formal clinical trials
tolerability of luspatercept - Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 52 weeks
  - To evaluate tolerability of luspatercept in subjects with transfusion-dependent beta thalassemia with baseline transfusion needs and comorbidities that were exclusion criteria in formal clinical trials
Efficacy of luspatercept - Number of subjects who showed a ≥ 33% reduction from baseline in the number of transfused blood units during any 12-week interval period of luspatercept treatment | 52 weeks
  - To evaluate efficacy of luspatercept in subjects with transfusion-dependent beta thalassemia with baseline transfusion needs and comorbidities that were exclusion criteria in formal clinical trials
impact of luspatercept on iron accumulation cardiac T2* | 52 weeks
  - To increase available data on the impact of luspatercept on iron accumulation by assessing the change in serum ferritin and cardiac T2* value on nuclear magnetic resonance imaging
impact of luspatercept on iron accumulation hepatic T2* | 52 weeks
  - To increase available data on the impact of luspatercept on iron accumulation by assessing the change in serum ferritin and hepatic T2* value on nuclear magnetic resonance imaging
incidence of endocrinological changes | 52 weeks
  - To evaluate the incidence of endocrinological changes in patients treated with luspatercept
incidence of thromboembolic events | 52 weeks
  - To assess the incidence of thromboembolic events in this category of patients
positively affect drug response. | 52 weeks
  - To identify the factors that positively affect drug response.
negatively affect drug response. | 52 weeks
  - To identify the factors that negatively affect drug response.

CONTACTS AND LOCATIONS:
Locations (1):
- UniversityCagliari, OspPed Microcitemico, Cagliari, Cagliari, Italia, Italy

IPD SHARING:
Plan to Share IPD: No